CLINICAL TRIAL: NCT02592967
Title: An Open Label Phase 1 Study of Safety and Immunogenicity of JNJ-64041757, A Live Attenuated Listeria Monocytogenes Immunotherapy, in Subjects With Non-Small Cell Lung Cancer
Brief Title: Safety & Immunogenicity of JNJ-64041757, Live-attenuated Double-deleted Listeria Immunotherapy, in Subjects With Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development of JNJ-64041757 discontinued due to lack of efficacy. No further follow up data will be collected after October 22, 2018.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107667; 64041757LUC1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; JNJ-64041757; Listeria monocytogenes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1A and 1B (Experimental): JNJ-64041757 will be administered intravenously (IV) once every 21 days.
  Interventions: Biological: JNJ-64041757 (Cohort 1A and 1B)
- Cohort 2A and 2B (Experimental): JNJ-64041757 will be administered intravenously (IV) once every 21 days.
  Interventions: Biological: JNJ-64041757 (Cohort 2A and 2B)

INTERVENTIONS:
Biological: JNJ-64041757 (Cohort 1A and 1B) — JNJ-64041757 will be administered IV at a lower dose in Cohort 1A (1x10^8 colony forming units [CFU] ) and at a higher dose in Cohort 1B (1x10^9 CFU)
  Arms: Cohort 1A and 1B
Biological: JNJ-64041757 (Cohort 2A and 2B) — JNJ-64041757 will be administered intravenously (IV) once every 21 days at the recommended dose as determined in Cohort 1A or 1B.
  Arms: Cohort 2A and 2B

SUMMARY:
The purpose of this study is to determine the recommended Phase 2 dose (RP2D) of JNJ-64041757 a live attenuated double deleted (LADD) Listeria monocytogenes (bacteria in which two virulence genes, which encode molecules that help cause disease, have been removed) when administered intravenously to participants with advanced (Stage IIIb) or metastatic (Stage IV) NSCLC (adenocarcinoma).

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1, open-label, multicenter and 2-part study in participants with advanced (Stage IIIb) or metastatic (Stage IV) non-small cell lung cancer (NSCLC) (adenocarcinoma). Part 1 of study will be Dose Escalation phase to determine the recommended Phase 2 dose (RP2D) based on safety and pharmacodynamic assessments and Part 2 will be Dose Expansion Phase to evaluate 2 expansion cohorts (Cohort 2A and 2B) after the RP2D for JNJ-64041757 is determined in Part 1. The study will consist of a Screening Period (from signing of informed consent until immediately before the first dose), an open-label Treatment Period (from the first dose of study drug until the End-of-Treatment Visit); and a Post treatment Follow-up Period (after the End-of Treatment Visit until study discontinuation). Dose limiting toxicity (DLT) in part 1, antigen-specific T-cell response in part 2 and incidence of adverse events in both the parts will be primarily evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Disease-related criteria for Part 1 and Part 2: 1) Histologically or cytologically documented non-small cell lung cancer (NSCLC) - adenocarcinoma; 2) Stage III b or IV disease; 3) Tested for presence of echinoderm microtubule-associated protein-like 4 anaplastic lymphoma kinase (EML4-ALK) rearrangement; 4) Received at least 2 prior lines of Food and Drug Administration (FDA)-approved systemic therapy, of which one therapy has to be a platinum-containing regimen OR failed or completed a first-line platinum-containing regimen and refused a second-line regimen despite being informed about the different therapeutic options and their specific clinical benefit by the investigator; the content of this informed consent discussion including the therapeutic options reviewed by the investigator needs to be documented and the subject needs to sign a specific consent form; Disease-related criteria for Cohort 2B only: 1) Mesothelin protein overexpression, defined by immunohistochemistry (IHC) as detection of the protein by greater than or equal (>=) 50 percent (%) of tumor cells on archived tumor material; 2) Primary tumor or metastatic lesion(s) amenable to tumor core biopsies
* At least 1 measurable tumor lesion per RECIST v1.1 (exception: subjects in Part 1 are not required to present with measurable disease)
* Eastern Cooperative Oncology Group (ECOG) Performance status score of 0 to 1
* At least 28 days since the last chemotherapy or immunotherapy prior to the first dose; at least 14 days since the last radiation prior to the first dose (exception: palliative radiotherapy for pain can be used greater than or equal to (>=) 7 days prior to or after infusion)

Exclusion Criteria:

* Untreated brain metastases. Subjects must have completed treatment for brain metastasis, and be neurologically stable off steroids, for at least 28 days prior to first dose of study drug
* History of listeriosis or vaccination with a listeria-based vaccine or prophylactic vaccine (eg, influenza, pneumococcal, diphtheria, tetanus, and pertussis [dTP/dTAP]) within 28 days of study treatment
* Known allergy to both penicillin and trimethoprim/sulfamethoxazole. Participants who are allergic to only one of these antibiotics are allowed to enroll
* Concurrent treatment with anti-Tumor necrosis factor alpha (TNF alpha) therapies, systemic corticosteroids (prednisone dose greater than [>]10 mg per day or equivalent) or other immune suppressive drugs within the 2 weeks prior to Screening. Steroids that are topical, inhaled, nasal (spray) or ophthalmic solution are permitted
* Positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of Dose-limiting toxicity (DLT) | First 21 days after the first infusion
  Percentage of participants who experienced DLT will be evaluated. The DLT dose level is defined as an unacceptable level of toxicity as evidenced by a DLT rate of greater than or equal to (>=) 33%.
Part 2: Antigen-specific T-cell Response | up to 1 year
  Biomarker analyses leukapheresis will be performed to evaluate immune responses to the vaccine after an single IV immunization.
Part 1 and Part 2: Incidence of Adverse Events (AEs) | From signing of informed consent form to 30 days after last dose of study drug
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; suspected transmission of any infectious agent via a medicinal product and medically important. Incidence was defined as the number of participants who experienced an adverse event within their period of participation in this study. Severity of adverse events will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE).

SECONDARY OUTCOMES:
Part 1 and Part 2: Objective Response Rate (ORR) | Baseline up to 30 days after last dose of study drug
  Objective response rate is defined as the percentage of participants who achieve complete response (CR) or partial response (PR), as assessed by the investigator.
Part 1 and Part 2: Duration of Response (DOR) | Baseline up to 30 days after last dose of study drug
  Duration of response will be calculated from the date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease (or relapse for subjects who experience CR during the study) or death.
Part 1 and Part 2: Progression-free Survival (PFS) | Baseline up to 30 days after last dose of study drug
  Progression-free survival is defined as the duration from the date of first dose of study drug until the date of first documented evidence of progressive disease (or relapse for subjects who experience CR during the study) or death, whichever comes first.
Part 1 and Part 2: Blood Culture Assessment of JNJ-64041757 | Periodically during treatment and up to one year after End of Treatment (EOT) visit
  This assessment will include the reporting of surveillance blood cultures (peripherally drawn, and through venous access device [if applicable]) for 1 year after the completion of JNJ-64041757 therapy.
Part 1 and Part 2: Shedding Profile of JNJ-64041757 From Cultured Samples of Feces, Urine, and Saliva | During cycle 1 (up to 21 days of treatment period) and at EOT visit (within 30 days after last dose)
  The shedding profile of JNJ-64041757 will be studied in cultures of (1) feces by stool or rectal swab, (2) urine samples, and (3) saliva samples.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (9):
- United States (9):
  - Duarte, California
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas

REFERENCES:
- [Background] Brockstedt DG, Giedlin MA, Leong ML, Bahjat KS, Gao Y, Luckett W, Liu W, Cook DN, Portnoy DA, Dubensky TW Jr. Listeria-based cancer vaccines that segregate immunogenicity from toxicity. Proc Natl Acad Sci U S A. 2004 Sep 21;101(38):13832-7. doi: 10.1073/pnas.0406035101. Epub 2004 Sep 13. PMID 15365184
- [Background] Le DT, Dubenksy TW Jr, Brockstedt DG. Clinical development of Listeria monocytogenes-based immunotherapies. Semin Oncol. 2012 Jun;39(3):311-22. doi: 10.1053/j.seminoncol.2012.02.008. PMID 22595054